CLINICAL TRIAL: NCT05795621
Title: A Multicenter, Randomized, Double-masked, Placebo-controlled Phase II/III Study Evaluating the Efficacy and Safety of IBI311 in Subjects With Active Thyroid Eye Disease
Brief Title: A Study of IBI311 in Subjects With Active Thyroid Eye Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI311A201
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants with TED will be randomized to receive 4 intravenous infusions of Placebo with an interval of 3 weeks for phase II and 8 intravenous infusions of Placebo with an interval of 3 weeks for phase III.
  Interventions: Biological: IBI311; Biological: placebo
- IBI311 (Active Comparator): Participants with TED will be randomized to receive 4/8 intravenous infusions of IBI311 with an interval of 3 weeks for phase II/III.
  Interventions: Biological: IBI311

INTERVENTIONS:
Biological: IBI311 — 10 mg/kg on Day 1 followed by 20 mg/kg q3W for the remaining 7 infusions for phase II/III.
Biological: placebo — 4 does of placebo for phase II; 8 does of placebo for phase III.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-masked, placebo-controlled Phase II/III study in subjects with active thyroid eye disease. Approximately 114 subjects meeting study eligibility criteria will be randomly assigned to IBI311 or placebo on day 1 (D1) in a 2:1 ratio stratified by smoking status

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent.
2. Male or female subject between the ages of 18 and 80 years, inclusive, at Screening.
3. Weight between 45 and 100 kg (inclusive).
4. Clinical diagnosis of Graves' disease associated with active TED with a CAS ≥ 3 for at least one eye at Screening and Baseline.
5. Moderate-severe active TED (not sight-threatening but has an appreciable impact on daily life), usually associated with at least two of the following: lid retraction ≥2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia.
6. Female Subjects should be fertile women who are sterile or have a negative blood pregnancy test during the screening period and who agree to take contraceptive measures within 120 days from the screening period to the last medication; Male subjects should agree to use contraception from the screening period to 120 days after the last dose.

Key Exclusion Criteria:

Subjects will be ineligible for study participation if they meet any of the following criteria:

1. At the time of screening, according to the subject's chief complaint or medical record, the time of first symptoms of active thyroid eye disease appeared in > 270 days;
2. Optimal corrected vision loss due to optic neuropathy, defined as two lines of vision loss due to optic neuropathy within the past 180 days, new visual field defects, or color vision impairment secondary to optic nerve involvement;
3. Corneal ulcers with no relief after treatment were determined by the investigator;
4. Baseline CAS decreased by more than 2 points compared with screening;
5. At any time prior to baseline or during the study period planned to receive orbital radiation therapy or TED specific surgery, including orbital decompression, strabismus surgery, and eyelid retraction correction;
6. Poor thyroid function control was defined as free triiodothyronine (FT3) or free tetriodothyronine (FT4) deviated more than 50% from the normal reference range of the local research center laboratory during screening;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
The proptosis responder rate of the study eye (defined as percentage of subjects with a ≥ 2mm reduction from Baseline in proptosis in the study eye, without deterioration [≥ 2 mm increase] of proptosis in the non-study eye). | Week 12 for phase II, Week 24 for phase III
  proptosis assessment: amount of protrusion of the eye from the orbital rim measured by Hertel exophthalmometer

SECONDARY OUTCOMES:
The overall responder rate in the study eye. | Week12 and Week24 for phase II, Week 24 for phase III
  Responder rate were defined as participants with a reduction in clinical activity score (CAS, see Secondary Outcome Measure 2 description for details) of ≥ 2 points, and a reduction in proptosis of ≥ 2 mm in the study eye, and no deterioration (increase in CAS of ≥ 2 points or increase in proptosis of ≥ 2 mm) in the non-study eye.)
Percentage of subjects with a CAS value of 0 or 1 in the study eye. | Week12 and Week24 for phase II, Week 24 for phase III
  According to the 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amendment, CAS was used to evaluate clinical activity. For each of the following items, one point is given:
  spontaneous orbital pain, gaze evoked orbital pain, eyelid swelling that is considered to be due to active (inflammatory phase) Graves' ophthalmopathy (GO), eyelid erythema, conjunctival redness that is considered to be due to active (inflammatory phase) GO, chemosis, and inflammation of caruncle or plica. The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity.
Mean Change of the CAS value in the study eye. | Baseline to Week 12 and Week 24 for phase II
Mean change from Baseline in proptosis measurement in the study eye. | Baseline to Week 12 and Week 24 for phase II, Baseline to Week 24 for phase III
  proptosis measurement: see Primary Outcome Measure 1 description for details
The proptosis responder rate of the study eye. | Week 24 for phase II
  proptosis responder rate: see Primary Outcome Measure 1 description for details
The diplopia responder rate of the study eye. | Week12 and Week24 for phase II, Week 24 for phase III

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Sun J, Li Y, Zhu L, Shan Z, Lu W, Shen J, Shi Y, Tao L, Jiang H, Ji L, Zhu Y, Gu H, Liu X, Sun B, Tian Y, Liu Q, Zhou J, Zhao H, Guan H, Zhu L, Wen J, Lu Y, Qiao J, Zhang W, Deng J, Lu S, Han-Zhang H, Qian L, Zhou H, Fan X. IGF-1R Inhibitor IBI311 for the Treatment of Active Thyroid Eye Disease in Chinese Patients: The RESTORE-1 Randomized Clinical Trial. JAMA Ophthalmol. 2025 Nov 1;143(11):964-971. doi: 10.1001/jamaophthalmol.2025.3350. PMID 41066129